CLINICAL TRIAL: NCT04326101
Title: Patient NT-proBNP Values and Medication Adherence on Their GP's Screen to Guide Dose Adjustment in Heart Failure (LabAdhDoc)
Brief Title: Electronic Transmission of Laboratory and Adherence Records of Heart Failure Patients to General Practitioners Screen
Acronym: LabAdhDoc
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01248
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transmission of adherence records — Electronic transmission of patient adherence records by pharmacists into medical EHR (Electronic Health Records)

SUMMARY:
Patients with heart failure (HF) need multiple guideline-directed medications to control the systolic and/or diastolic ventricular dysfunction. Laboratory measure the biomarker NT-proBNP (N-terminal pro-B type natriuretic peptide) to support clinical decision and to guide treatment at every stage of HF. Many patients (including HF patients) do not follow therapeutic recommendations. Electronic monitoring of medication intake gives precise information over time and is the gold standard to unveil inappropriate behaviour. Electronic Health Records (EHR) are repository of patient health data in digital format and are mostly locally configured in medical practices.

We aim to transmit laboratory results of NT-proBNP and estimates of medication adherence into the EHR system of primary care providers, with the objective to guide treatment and dose adjustment of multiple medications in patients with HF. Our project is *not* to develop a telemonitoring system.

DETAILED DESCRIPTION:
Patients with heart failure (HF) need multiple guideline-directed medications to control the systolic and/or diastolic ventricular dysfunction. To support clinical decision and to guide treatment at every stage of HF, the measurement of the biomarker NT-proBNP (N-terminal pro-B type natriuretic peptide) has been recommended.

Many patients (including HF patients) do not follow therapeutic recommendations. Non-adherence to treatment can lead to acute decompensation that often requires urgent hospitalisation. Electronic monitoring of medication intake gives precise information over time and is the gold standard to unveil inappropriate behaviour. We developed Time4MedTM, a small device that records date and time of medication intake. The recorded electronic data are visualized in a scatter diagram and several adherence estimates can be calculated such as days with missed doses, taking adherence or timing adherence. Electronic Health Records (EHR) are repository of patient health data in digital format and are mostly locally configured in medical practices.

We aim to transmit laboratory results of NT-proBNP and estimates of medication adherence into the EHR system of primary care providers, with the objective to guide treatment and dose adjustment of multiple medications in patients with HF. Our project is *not* to develop a telemonitoring system.

This is a prospective, observational, feasibility study one medical practice in Basel-Stadt, one dedicated laboratory, and one community pharmacy as study centre.

Physicians will order NT-proBNP measurement and electronic adherence monitoring to patients with diagnosis New York Heart Association (NYHA) stage II-III, who are under guidelines-recommended multiple medications and whose clinical and/or biomedical targeted values are unmet (inadequate control). Laboratory and adherence reports will be generated in similar encrypted format and transferred via secured platform into physician's EHR.

We expect to show that electronic adherence reports can be gathered and electronically transferred by pharmacists into medical EHR in the same way as laboratory reports. The joint availability of medication adherence estimates and laboratory values in the EHR can guide physicians in the management and therapy of patients with HF.

ELIGIBILITY:
Inclusion Criteria:

* is ≥ 18 years old;
* was diagnosed with HF NYHA II-III;
* is under multiple regimen (ACE-Inhibitors and/or mineralocorticoid receptor antagonist (MRA) and/or betablocker (BB) and/or diuretic and/or other);
* did not reach targeted clinical and/or biomedical objectives (HF is inadequately controlled);
* self-administers medication (no help or supervision from a third person);
* is suspected of inappropriate intake behaviour;
* accepts to use the monitoring device for one month;
* accepts a home-visit from the study pharmacist one month later;
* signs the informed consent form.

Exclusion Criteria:

- Patients who are, in the opinion of the physician, unlikely to comply with the study schedule or are unsuitable for any other reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: suffers from heart failure NYHA II-III
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Successful transmission | one month
  The adherence records transmitted by the pharmacy are available in the health records system of GPs

SECONDARY OUTCOMES:
Physician satisfaction | through study completion, 1 year
  Satisfaction of physician with the availability of adherence records in his/her health records system

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof, Study Chair — University of Basel
Locations (1):
- Praxis Hammer, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dietrich F, Zeller A, Allemann S, Arnet I. Development and acceptance of a new adherence monitoring package to identify non-adherent patients with polypharmacy in primary care: a feasibility study. BMJ Open Qual. 2023 Feb;12(1):e002155. doi: 10.1136/bmjoq-2022-002155. PMID 36849193